CLINICAL TRIAL: NCT03340389
Title: Dysfunctional Lens Index Serves as a Novel Surgery Decision Maker for Age-related Cataracts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, yin ying zhao, Director, Wenzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: DLI_HZ
Record Dates: First submitted 2017-11-06; First posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Age-related Cataract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cataract surgery (Experimental): cataract extraction and intraocular implantation
  Interventions: Procedure: a ray-tracing aberrometry

INTERVENTIONS:
Procedure: a ray-tracing aberrometry — The Dysfunctional Lens Index is obtained by a ray-tracing aberrometry

SUMMARY:
To study the correlations among the dysfunctional lens index (DLI), Lens Opacities Classification System III (LOCS III) nuclear opalescence grading score, preoperative corrected distance visual acuity (CDVA), the objective scatter index (OSI) and Scheimpflug based average lens density in age-related cataracts. To investigate the potential of the DLI as a novel surgery decision maker via the Operating Characteristic (ROC) curve analysis.

DETAILED DESCRIPTION:
Each patient received a comprehensive eye examination, including corrected distance visual acuity (CDVA) preoperatively and the day after surgery, subjective refraction, slit-lamp evaluation, noncontact tonometry (TX-F; Cannon, Tokyo, Japan), and dilated fundus examination. According to the surgery decision made by the three surgeons based on the slit lamp biomicroscopy and CDVA, patients were divided into two groups: Surgical and Non-Surgical. The results of the DLI, OSI and average lens density (ALD) were masked to the surgeons. The DLI, OSI, average lens density, LOCS III nuclear opalescence grading, and preoperative CDVA were obtained. Correlations among these parameters were analyzed. ROC curves were used to analyze DLI values to determine a value to separate between surgical and non-surgical cataracts.

ELIGIBILITY:
Inclusion Criteria:

* patients with age-related cataracts

Exclusion Criteria:

* any corneal opacity, corneal dystrophies, retinal anomalies, a history of ocular surgery or laser treatment, a LOCS III grade of cortical opacity ≥ 3.0 or posterior subcapsular cataract ≥ 2.0.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-05-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Dysfunctional lens index | 6 months
  The DLI is an objective lens performance metric derived from internal higher order aberrations (HOAs), pupil size, and contrast sensitivity data

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No